CLINICAL TRIAL: NCT00733382
Title: The Effect of Dexamethasone in the Attack of Migraine Headache and to Prevent of Its Relapse After Discharge From Emergency Department: a Randomized, Double-Blind, Controlled Trial.
Brief Title: Effect of Dexamethasone on Migraine Headache
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Shiraz University of Medical Sciences (Other)
Responsible Party: Reza Nemati/research manager of neurology department, Shiraz university of medical sciences
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: 212110
Record Dates: First submitted 2008-08-11; First posted 2008-08-13 (Estimated); Last update posted 2008-08-13 (Estimated); Status verified 2008-08

CONDITIONS: Migraine Headache
Keywords: migraine; dexamethasone; dihydroergotamine
MeSH Terms: conditions — Migraine Disorders | interventions — 21-benzyloxy-9alpha-fluoro-16alpha-methylpregna-1,4-dien-11beta,17alpha-diol-3,20-dione

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental)
  Interventions: Drug: dexamethazone
- 2 (Active Comparator)
  Interventions: Drug: dexamethazone

INTERVENTIONS:
Drug: dexamethazone — injection form, 8 miligram, injected once

SUMMARY:
Dexamethasone is a safe and cheap abortive therapy for migraine headache. The effect of it is never evaluate and not correlate with the effect of popular anti migraine medication such as dihydroergotamine. The investigators proposal is to compare its effect with dihydroergotamine.

ELIGIBILITY:
Inclusion Criteria:

1. Migraine attack according to international headache society criteria
2. Migraine without aura; at least 5 attack with mean duration of 4 to 72 hours and 2 of following:

   * Unilateral
   * Pulsatile
   * Severe enough to impair daily activity
   * Aggravate with walking and climbing, also 1 of following:

     * Nausea and or vomiting
     * Photophobia and phonophobia, and not contributed to other headache.
3. Migraine with aura; at least 2 attacks with 3 of following:

   * One reversible aura
   * Aura became apparent at least in 4 minutes
   * Aura not lasting more than 60 minutes
   * Headache develops in less than 60 minutes after aura

Exclusion Criteria:

1. Hypertension
2. Ischemic heart disease
3. Basilar migraine with sign and symptoms such as:

   * Diplopia
   * Ataxia
   * Dysarthria
   * Dysphagia
   * Weakness
   * Sensory disorder
   * Drowsiness
4. Peripheral vascular disease
5. Sepsis
6. Age more than 40 and less than 15 year old
7. Pregnancy
8. Use of triptans and ergots derivatives in past 24 hours

Ages: 15 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 30 (Estimated)
Dates: Start 2008-02; Primary Completion 2008-12 (Estimated); Study Completion 2009-08 (Estimated)

PRIMARY OUTCOMES:
to evaluate the efficacy of dexamethazone in abortive therapy of migraine attack and prevent of recurrence

CONTACTS AND LOCATIONS:
Locations (1):
- Peyman Petramfar, Shiraz, Fars, Iran